CLINICAL TRIAL: NCT02792608
Title: A Mindfulness-Based Intervention to Improve Quality of Life Among Brain Tumour Survivors
Brief Title: Mindfulness-Based Therapy for Brain Tumour Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Brain Tumour Foundation of Canada (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 169-2015
Record Dates: First submitted 2016-05-26; First posted 2016-06-07 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2018-06

CONDITIONS: Brain Tumour; Depressive Symptoms; Survivors
Keywords: Mindfulness-based Therapy; Brain Tumour Survivors; Depressive Symptoms; Quality of Life; Perceived Stress; Wellbeing; Treatment
MeSH Terms: conditions — Brain Neoplasms; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness-based Therapy (Experimental): 5 week, manual-based group MBI treatment for depression
  Interventions: Behavioral: Mindfulness-based Therapy

INTERVENTIONS:
Behavioral: Mindfulness-based Therapy — MBT will be delivered in group format, 135 minutes per week, for 5 consecutive weeks with 10-20 participants per group.

SUMMARY:
Brain Tumour (BT) survivors struggle with disabling physical, emotional, cognitive and psychosocial sequelae. Unfortunately, to-date there has been very limited research into rehabilitative interventions for this population. With 55,000 BT survivors in Canada alone1, access to effective, evidence-based rehabilitative treatment that would improve BT survivors' quality of life (QOL) and capacity to cope is a necessity. Mindfulness-Based Therapy's (MBTs) are emerging as a potential treatment to address this need. MBTs are group-based psychological treatments for coping with illness or disability, with the goal of improving psychological wellbeing. Recent studies have begun to suggest a role for MBTs in addressing symptom burden and QOL in the acquired brain injury (ABI) population, a heterogeneous population that includes survivors of stroke and traumatic brain injury, as well as BT survivors. High quality research including within-subject controlled trials, are needed to demonstrate whether MBTs can provide efficacious, accessible and cost-effective treatment to improve the lives of BT survivors.

DETAILED DESCRIPTION:
Increased survival rates and life expectancy of primary BT survivors today have resulted in a need to expand the focus from acute treatment to reducing disability and long-term symptom burden in survivorship. Many BT survivors are left with reduced autonomy in their lives, with a lower likelihood of independent living and increased risk of functional and symptom adversity (pain and physical disability), unemployment, and family difficulties. Unsurprisingly, these factors are associated with increased stress, psychological suffering, and reduced QOL. Research has noted the prevalence of psychological distress and cognitive impairment, experienced as late effects, with up to 90% of survivors experiencing some form of cognitive impairment and depressive symptoms, as well as many as 80% experiencing mental fatigue and up to 60% experiencing anxiety.

80% of all central nervous system tumour survivors exhibit rehabilitation needs, and survivors report an interest in learning coping techniques for stress, yet the majority of symptoms remain underestimated and untreated. BT survivors are left with limited treatment options to promote long-term wellbeing, with 71% of resources containing minimal to no information on coping with outcomes. Despite considerable research demonstrating BT survivors increased risk of symptom burden and reduced QOL, there has been little research on treatment or effective interventions.

Some outpatient rehabilitation therapies have been made available to other neurologically impaired populations (e.g. Traumatic Brain Injury, Stroke) but evidence in support of specific approaches has been equivocal, with limited rehabilitative research in BT survivors specifically. Such treatments for the broader ABI population to-date have included Cognitive Behavioural Therapy (CBT) and Applied Behavioural Analysis (ABA), with debatable effectiveness. Positive studies have suggested that treatment may only prove effective for a handful of ABI sequelae. Studies to date are marred by limited methodological rigour and applicability to the BT population because of the broader, heterogeneous ABI focus. As a result, healthcare professionals and national organizations, such as National Coalition for Cancer Survivorship, have called for higher quality research to inform novel treatments to improve outcomes for specific groups, such as the BT population.

In response to these calls, Mindfulness-Based Therapy's (MBTs) have been proposed as a plausible treatment for long term care of ABI survivors, in general. MBTs use a non-stigmatizing approach, combining secularized eastern meditative practices with western psychological advances. MBTs have good evidence that they improve a wide range of sequelae, including, stress, depression, anxiety and cognitive impairment. MBT efficacy has been repeatedly demonstrated across multiple psychiatric, neurological, and cancer populations. MBTs focus on acceptance-based and adaptive approaches, which might theoretically be better suited to the realities of the lives of BT survivors, than would change-based approaches such as CBT or ABA. MBT participants learn to generate less distress, engage more positively in their lives, and respond to difficult situations more adaptively; they often describe it as transformative.

MBTs have begun to be studied in the broader ABI survivor population, and this emerging literature suggests efficacy in reducing symptom burden. However, there are no known studies considering the effectiveness of an MBT for BT survivors specifically; the present study aims to fill this important knowledge gap. The goal of this study is to test the effectiveness of a five session MBT course in reducing depressive symptoms and perceived stress, as well as improving overall QOL and wellbeing for BT survivors.

ELIGIBILITY:
Inclusion Criteria:

* consenting brain tumour survivor at The Odette Cancer Centre
* >six months post-treatment
* Ability to communicate, in written and spoken English

Exclusion Criteria:

* Minimal depressive symptoms (score below 14 on the BDI-II)
* Previous head injuries or non-BT neurological diseases
* Unaware of deficits (determined through clinical judgement)
* Substance abuse / dependence within three months
* History of dementia, a recent suicide attempt, or current self-injurious behavior
* Previously completed >four weeks of a MBI, or general CBT, in the past three years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Depressive Symptoms at 5 Weeks | Pre- (Week 0) and Post-Treatment Assessment (Week 5)
  Scale used to measure Depressive Symptoms: Beck Depression Inventory II (BDI-II)

SECONDARY OUTCOMES:
Change from Baseline Quality of Life at 5 Weeks | Pre- (Week 0) and Post-Treatment Assessment (Week 5)
  Scale used to measure Quality of Life: Quality of Life after Brain Injury (QOLBRI)
Change from Baseline Perceived Stress at 5 Weeks | Pre- (Week 0) and Post-Treatment Assessment (Week 5)
  Scale used to measure Perceived Stress: Perceived Stress Scale (PSS)
Change from Baseline Mental Wellbeing at 5 Weeks | Pre- (Week 0) and Post-Treatment Assessment (Week 5)
  Scale used to measure Mental Wellbeing: Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Selchen, MD MSt FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre; Janet Ellis, MB MD FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No